CLINICAL TRIAL: NCT05935007
Title: Aveir Dual-Chamber Leadless Pacemaker Real-World Evidence Post-Approval Study
Brief Title: Aveir DR Real-World Evidence Post-Approval Study
Status: Recruiting | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: ABT-CIP-10454
Record Dates: First submitted 2023-05-24; First posted 2023-07-07 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Cardiac Pacemaker; Arrythmia; Bradycardia
Keywords: bradycardia; sick sinus rhythm; pacemaker; av block; vasovagal syncope
MeSH Terms: conditions — Arrhythmias, Cardiac; Bradycardia; Atrioventricular Block; Syncope, Vasovagal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Interventions: Device: Aveir DR Leadless Pacemaker System
  This study will utilize real-world data from patients implanted with the Aveir DR Leadless Pacemaker System. No device intervention will be conducted in this study.
  Interventions: Device: Aveir DR Leadless Pacemaker System

INTERVENTIONS:
Device: Aveir DR Leadless Pacemaker System — This study will utilize real-world data from patients implanted with the Aveir DR Leadless Pacemaker System. No device intervention will be conducted in this study.

SUMMARY:
The purpose of this post-approval study is to evaluate the long-term safety of the dual-chamber Aveir DR leadless pacemaker using real-world evidence methods.

DETAILED DESCRIPTION:
This is a non-randomized, multi-center study leveraging real-world evidence methods that merge multiple real-world datasets from Abbott and the Center for Medicare Services to assess Aveir DR leadless pacemaker safety in a large patient population. The results from this study will provide long-term safety data for the Aveir dual chamber LP and the Aveir atrial LP to fulfill the Condition of Approval requirements for the Aveir DR device from FDA.

Due to the RWE data collection methods used in this study, a central IRB approved informed consent waiver has been granted. Due to this waiver and the sponsor's use of the central IRB, individual hospitals are not required to consent patients or complete local IRB submissions for this RWE study.

ELIGIBILITY:
Eligibility Criteria:

* Implanted with an Aveir DR leadless pacemaker
* Continuous enrollment in Medicare Part A and Part B for 12 months prior to implant and for -30 days after implant, except in the case of death within the 30-day period
* Ability to link with Medicare fee-for-service data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who had an implant of the Aveir DR device, meet inclusion/exclusion criteria, link to Medicare FFS claims, and survive past 30 days will be included in the analysis
Sampling Method: Probability Sample
Enrollment: 1805 (Estimated)
Dates: Start 2023-10-31 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Number of Subjects Free from Acute Aveir DR System-Related Complications | 30 Days
  Freedom from key acute complications through 30 days post implant procedure
Number of Subjects Free from Chronic Aveir DR System-Related Complications | 5 Years
  Freedom from key chronic complications from 31 days through 5 years post implant procedure procedure

SECONDARY OUTCOMES:
Number of Subjects Free from Individual Aveir DR Leadless Pacemaker-Related | 5 Years
  Complication rate of the Aveir DR leadless pacemaker for key individual acute and chronic complications
Number of Subjects with End of Device Service Events | 5 Years
  Care of subjects at the end of device service. End-of-device service is defined as any event prior to the 5-year follow-up period which results in the leadless pacemaker being explanted or deactivated, another CIED implanted, or death. All instances of the end-of-service will be summarized by event type and time to event.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Harbert, Study Director — Abbott
Locations (1):
- Abbott, Sylmar, California, United States

IPD SHARING:
Plan to Share IPD: No